CLINICAL TRIAL: NCT05498740
Title: Post-marketing Study in Femoral Popliteal Artery of Drug Coated Ballon Used for Treatment of Lower Limb Ischemia
Brief Title: Post-marketing Study in Femoral Popliteal Artery of Drug Coated Balloon Used for Treatment of Lower Limb Ischemia
Acronym: UltraFuture I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04202106
Record Dates: First submitted 2022-07-22; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- drug eluting balloon catheter (Experimental): use drug eluting balloon catheter to treat the stenosis or occlusion in superficial femoral artery(SFA) and/or popliteal artery
  Interventions: Device: Drug eluting Balloon

INTERVENTIONS:
Device: Drug eluting Balloon — Drug eluting Balloon is a kind of the product that has been used for many years. By filling the micropores on the surface of the balloon with anti-proliferative drugs like immunosuppressive agents, the balloon is expanded and contacted with the lesion to rapidly release the drug to the local arterial wall.

SUMMARY:
The objective of this prospective, multi-center, single arm study is to obtain further data on the safety and performance of the Drug-coated Balloon catheters in the treatment of the Superficial Femoral Artery (SFA) and Popliteal Arteries (PA).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤85 years old
2. Rutherford clinical category classification：2-5
3. Significant stenosis (≥50%) or occlusions of lesion(s) located in the superficial femoral artery an /or the popliteal artery
4. At least one patent native outflow artery to the ankle free from significant lesion as confirmed by angiography
5. Subject has provided written informed consent prior to participation , understands the purpose of this trail and agrees to comply with all protocol-specified examinations and follow-up appointments.

Exclusion Criteria:

1. Aneurysms near target lesions or popliteal aneurysms.
2. The guide wire cannot pass smoothly through the target lesion.
3. Known allergy to contrast agents, heparin or paclitaxel.
4. Patient already enrolled in other investigational (interventional) studies that would interfere with study endpoints or may enroll in other studies after enrollment in this clinical trial.
5. Pregnancy or female patient with child bearing potential not taking adequate contraceptives or currently lactating.
6. Other comorbidities, which in the opinion of the investigator limit longevity or likelihood of compliance with protocol follow up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
rate of device success | intraoperative
rate of procedural success | intraoperative
rate of technical success | intraoperative
rate of primary patency of target lesion | 12 months
rate of primary patency of target lesion | 24 months
rate of Clinically-driven TLR | 12 months
rate of Clinically-driven TLR | 24 months
rate of TLR | 1 month
rate of TLR | 12 months
rate of TLR | 24 months
rate of Clinically-driven TVR | 12 months
rate of Clinically-driven TVR | 24 months
rate of TVR | 1 month
rate of TVR | 12 months
rate of TVR | 24 months
change in Rutherford clinical category (target limb) | 12 months
change in Rutherford clinical category (target limb) | 24 months
change in ankle brachial index(ABI) | 12 months
change in ankle brachial index(ABI) | 24 months
rate of SAE | 12 months
rate of SAE | 24 months
rate of All-cause mortality | 1 month
rate of All-cause mortality | 12 months
rate of All-cause mortality | 24 months
rate of Major amputation | 1 month
rate of Major amputation | 12 months
rate of Major amputation | 24 months
rate of target lesion thrombosis | 12 months
rate of target lesion thrombosis | 24 months
Rate of adverse events | intraoperative
Rate of adverse events | 1 month
Rate of adverse events | 12 months
Rate of adverse events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Fu, Principal Investigator — Shanghai Zhongshan Hospital
Locations (24):
- China (24):
  - Xuanwu hospital, Beijing
  - Affiliated Hospital of Chengde Medical College, Chengde
  - The Third People's Hospital of Chengdu, Chengdu
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - Guangzhou Huaqiao hospital, Guangzhou
  - Hospital of Traditional Chinese Medicine affiliated to Guangzhou Medical University, Guangzhou
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Ha’erbin
  - First Hospital of Lanzhou University, Lanzhou
  - Ningbo huamei hospital, Ningbo
  - Qingdao Municipal Hospital, Qingdao
  - Ruian People's Hospital, Rui’an
  - Shanghai Ninth People'S Hospital, Shanghai
  - Zhongshan Hospital, Shanghai
  - Northern Theatre General Hospital, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin People's Hospital, Tianjin
  - Weifang People's Hospital, Weifang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The First Affiliated Hospital of Xi 'an Jiaotong University School of Medicine, Xi'an
  - People's Hospital of Xinjiang Uygur Autonomous Region, Xinjiang

IPD SHARING:
Plan to Share IPD: No